CLINICAL TRIAL: NCT05383092
Title: Adapted Physical Activity for Children Treated With Cancer and Insulin Sensitivity
Acronym: APACIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/22/0061
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pediatric Cancer
Keywords: pediatric cancers; exercise; insulin sensibility; metabolic syndrome
MeSH Terms: conditions — Neoplasms; Motor Activity; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective randomized pilot study studying the parameters of two groups receiving physical activity management over a period of 6 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted physical activity Strong (Experimental)
  Interventions: Other: Adapted Physical Activity Strong
- Adapted physical activity Soft (Active Comparator)
  Interventions: Other: Adapted Physical Activity Strong

INTERVENTIONS:
Other: Adapted Physical Activity Strong — Children will practice physical activities combining aerobics and muscle strengthening. They will follow a 30-minute (for prepubescent children) or 60-minute (for pubescent children) Strong adapted physical activity session 2 to 3 times a week during hospitalization periods or by videoconference at home when they are not hospitalized.

SUMMARY:
The main objective of this study is to evaluate the evolution of the sensitivity to insulin, a hormone that acts on sugar in the body, as well as other metabolic, motor and nutritional elements of children with cancer, according to the practice of intense physical activities or stretching. In view of the scientific work on this subject, it is expect to observe that the practice of intense physical activities will improve the results of the children in the metabolic, motor and nutritional evaluations, compared to the stretching program.

DETAILED DESCRIPTION:
The protocol consists of 6 months of intense physical activity and stretching programs for children with solid cancer or haematological disease, starting at diagnosis. Evaluations will be performed at the first, third and sixth month of the programs and then six and eighteen months after they are stopped. The physical activity sessions will take place in the hospital during hospitalizations or by videoconference when the children are at home. The sessions are adapted to the needs, desires and abilities of the children and will take place two to three times a week. They will be mediated by various activities such as soccer, rugby, darts, muscle strengthening. Inclusion lasts two years.

ELIGIBILITY:
Inclusion Criteria:

* age between 5 and 18 years old;
* have a solid cancer or hematological disease;
* be treated for the first time in pediatric oncology and hematology department;
* have an estimated life expectancy at diagnosis of more than 6 months.

Exclusion Criteria:

* present a physical and/or psychological impossibility to follow an adapted physical activity program;
* have a pre-existing heart disease that is not suitable for adapted physical activities;
* have a known type 1 diabetes
* have an obesity defined by a body mass index greater than or equal to the International Obesity Task Force 25 threshold

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin Sensitivity | 6 months
  Homeostasis Model Assessment of Insulin Resistance

CONTACTS AND LOCATIONS:
Overall Officials: Marlène PASQUET, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- PASQUET Marlène, Toulouse, France

REFERENCES:
- [Derived] Thomas J, Filleron T, Auriol F, Laurens C, Pasquet M. Study protocol of an early randomized intervention trial assessing the metabolic effects of two levels of exercise intensity in children undergoing cancer treatment: the APACIS study. BMC Cancer. 2025 May 9;25(1):850. doi: 10.1186/s12885-025-14235-4. PMID 40346598